CLINICAL TRIAL: NCT00666432
Title: Bipolar and Schizophrenia Consortium for Parsing Intermediate Phenotypes
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, MPRC, L.E. Hong, University of Maryland, Baltimore
Other Study IDs: HP-00043960; R01MH077852 (NIH)
Record Dates: First submitted 2008-04-21; First posted 2008-04-24 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia; Bipolar
Keywords: schizophrenia; bipolar; eye movements; phenotype; biochemical; relatives
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood or saliva will be stored for future genetic analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Controls
  Interventions: Other: This is an observational study model that is family based
- 2: Patient Family
  Interventions: Other: This is an observational study model that is family based
- 3: Patients
  Interventions: Other: This is an observational study model that is family based

INTERVENTIONS:
Other: This is an observational study model that is family based — This is an observational study model that is family based

SUMMARY:
Briefly, this multisite study is designed to identify endophenotypes (i.e., heritable biomarkers) associated with either schizophrenia or bipolar disorder alone, or both together. The subsequent genetic analyses will search genomic loci and candidate genes associated with each of the independent endophenotypes. This is a five site study that is slotted for NIMH funding.

DETAILED DESCRIPTION:
We propose to recruit 100 case probands with a diagnosis of SZ, 100 case probands with a diagnosis of BP Disorder I with history of psychosis; BPI-P) and 400 1st degree case relatives. All 1st degree family members who are willing to participate will provide clinical information and blood sample, only a proportion will be eligible for endophenotypic studies). Individuals with psychotic disorder not otherwise specified are also eligible for testing. Their data will be incorporated with the schizophrenia or bipolar data upon confirmation of diagnosis. Family members of individuals with psychotic disorder not otherwise specified will not be tested unless the individual has a later confirmed diagnosis of schizophrenia or bipolar disorder. Probands will not be tested during the acute phase of the illness as judged clinically e.g., significant increase in core symptoms from their stable baseline that requires a change in treatment such increased dose of medication, drug change, or hospitalization). As part of another existing protocol, we have collected most of the endophynotypic information in schizophrenia probands and 1st degree relatives other than brain imaging and few other tests. We will attempt to recruit these subjects to complete the imaging studies and the data will be used in the current study.

We will recruit 100 healthy comparison subjects from the community in order to describe the distribution of normal values for our endophenotype procedures in a demographically matched sample. The SZ and BPI-P probands, and 50 healthy control subjects, will be frequency matched on age, sex ratio, and head of the household's socio-economic status (SES). Another group of 50 healthy control subjects will be similarly matched to the relative groups recruited.

Participants will undergo a number of clinical, electrophysiological, structural brain imaging, perceptual, and cognitive assessments. These data will be used to identify phenotypes likely to be associated with genetic risk for schizophrenia and/or bipolar disorder, and to determine how these phenotypes aggregate in families. Some of the analyses will focus on examining associations between candidate genes and these alternative phenotypes. Thus if we are not able to recruit relatives we may still collect these phenotypic data in probands and their genetic sample for future genotype/phenotype association studies. Family members may elect to participate only in the clinical and blood draw portions of the study. Testing procedures require a 12 -15 hour time commitment and testing will be completed over 2 or more days. Participants will be asked to give a blood (or saliva if difficult to obtain blood sample for instance because of fear of blood draws), which will be stored for future genetic analyses. Data from the previous family study will be combined with the data collected in this protocol for some of the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 15 years of age and above.
* Case probands will include individuals who meet DSM-IV criteria for schizophrenia, schizoaffective, or bipolar disorder with psychosis

Exclusion Criteria:

* Control subjects who meet DSM-IV criteria for any lifetime psychotic illness or BP, or have a family history of psychotic or BP disorders in their first or second-degree relatives will be excluded.
* A number of exclusions are necessary because they potentially affect neurophysiological measures. Exclusions will be applied to all groups to maintain consistency in recruitment. As a result, the following individuals will be excluded:
* Subjects under 15 years of age will be excluded. Subjects with serious medical, neuro-ophthalmological or neurological illness (e.g., cancer, seizure disorders, encephalopathy) will be excluded, with the exception of family member subjects participating for clinical interview and blood sample only.
* Subjects with current substance abuse (within 6 months), dependence within 2 years or extensive history of drug dependence will be excluded, with the exception of family member subjects participating for clinical interview and blood sample only.
* Subjects with mental retardation will be excluded, with the exception of family member subjects participating for clinical interview and blood sample only.
* Subjects with ferromagnetic objects lodged in body will be excluded, with the exception of family member subjects participating for clinical interview and blood sample only.
* Schizophrenic patients who are judged to be incompetent to provide voluntary informed consent based on the ESC evaluation.
* Any participant who would require an x-ray to rule out the presence of metal in their body prior to an MRI scan

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from the University of Maryland, Community Mental Health Center and Private Psychiatrists.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2008-05; Primary Completion 2012-09 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Smooth pursuit eye movement measures; P50 gating; PPI; Cognitive measures; P300 component of evoked potential; genetic markers | 10-13 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Liyi E Hong, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (6):
- United States (6):
  - Hartford Hospital- The Institute of Living, Hartford, Connecticut
  - Center for Cognitive Medicine, Chicago, Illinois
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Wayne State University School of Medicine, Detroit, Michigan
  - University of Texas Southwestern Medical Center, Dallas, Texas